CLINICAL TRIAL: NCT01590459
Title: A 24-week, Double-Blind, Randomized, Parallel Group, Placebo-Controlled, Phase 2 Study of Different Doses of VX-509 in Adult Subjects With Active Rheumatoid Arthritis on Stable Methotrexate Therapy With 104-Week Open Label Extension
Brief Title: 24-week Study With Open Label Extension of VX-509, an Oral JAK3 Inhibitor, in Subjects Taking Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX11-509-102; 2011-004419-22 (EudraCT Number)
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 2-((2-(1H-pyrrolo(2,3-b)pyridin-3-yl)pyrimidin-4-yl)amino)-2-methyl-N-(2,2,2-trifluoroethyl)butanamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: VX-509 matching placebo
- VX-509 100 mg qd Arm (Experimental)
  Interventions: Drug: VX-509
- VX-509 150 mg qd Arm (Experimental)
  Interventions: Drug: VX-509
- VX-509 100 mg bid Arm (Experimental)
  Interventions: Drug: VX-509
- VX-509 200 mg qd Arm (Experimental)
  Interventions: Drug: VX-509

INTERVENTIONS:
Drug: VX-509 — 50 mg oral tablet
  Arms: VX-509 100 mg bid Arm; VX-509 100 mg qd Arm; VX-509 150 mg qd Arm; VX-509 200 mg qd Arm
Drug: VX-509 matching placebo — 0 mg oral tablet
  Arms: Placebo Arm

SUMMARY:
This study is designed to evaluate the safety and efficacy of VX-509, an oral JAK3 inhibitor, for treatment of subjects with active RA who have had an inadequate response to Methotrexate.

DETAILED DESCRIPTION:
VX-509 is an oral, selective Janus kinase 3 (JAK3) inhibitor being developed by Vertex. In autoimmune diseases, JAK3 is an essential component of the immune signaling cascade. This cascade ultimately contributes to abnormal immune response that results in chronic inflammation and, in the case of rheumatoid arthritis (RA), irreversible damage to cartilage and bones. Selective inhibition of JAK3 offers a new disease modifying approach to the treatment of RA, and a broad range of other autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, between 18 and 80 years of age (inclusive)
* All subjects must have been diagnosed with RA
* Must have a swollen joint count of ≥6 out of 66 joints and tender joint count of ≥6 out of 68 joints
* Baseline CRP level must be above the upper limit of normal
* All subjects must have been receiving stable MTX coadministered with folic or folinic acid (at least 5 mg/week)
* Subjects may remain on 1 nonsteroidal anti-inflammatory medication during the study (aspirin ≤ 325 mg/day is allowed).
* Subjects must not have received prior treatment with a JAK inhibitor
* Subjects who are on an additional nonbiologic DMARD (e.g., sulfasalazine) must be willing to discontinue that DMARD after signing consent, except for hydroxychloroquine
* Subjects may have received previous therapy with a single TNF inhibitor (e.g., etanercept, adalimumab, infliximab, golimumab, certolizumab pegol)
* Females must have a negative pregnancy test prior to study dosing
* Sexually active subjects and their partners must agree to contraceptive requirements

Exclusion Criteria:

* History or presence of a clinically significant medical disorder other than RA that, in the opinion of the investigator and medical monitor, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Subjects with inflammatory, rheumatological disorders other than RA
* Pregnant or nursing female subjects
* Subjects who have a female partner who is pregnant, nursing, or planning to become pregnant
* Subjects who have planned major surgery (e.g., joint replacement) or procedures during the study
* History of drug abuse or positive drug screen
* History of alcohol abuse or excessive alcohol consumption
* History of tuberculosis (TB) infection of any kind (pulmonary or extrapulmonary, active or latent), regardless of history of anti-TB treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a 20% improvement in disease severity according to the American College of Rheumatology criteria, assessed using the C-reactive protein level (ACR20-CRP) response | Week 12
Change from baseline in Disease Activity Score 28 using C-reactive protein (DAS28- CRP) | Week 12
Safety and tolerability | Week 12
  Measured by incidence of treatment-emergent adverse events
Safety and tolerability | Week 12
  Measured by clinical laboratory values (serum chemistry, hematology, coagulation studies, and urinalysis)
Safety and tolerability | Week 12
  Measured by 12-lead ECG outcomes
Safety and tolerability | Week 12
  Measured by vital signs

SECONDARY OUTCOMES:
Proportion of subjects who achieve an ACR20-CRP response | Week 24
Proportion of subjects who achieve ACR50-CRP and ACR70-CRP responses | Week 12 and 24
Proportion of subjects who achieve a moderate or good response according to the European League Against Rheumatism (EULAR) response criteria | Week 12 and 24
Proportion of subjects who achieve remission as defined by DAS28-CRP response | Week 12 and 24
Proportion of subjects who achieve remission as defined by the ACR/EULAR definition of remission | Week 12 and 24
Change from baseline in selected Patient Reported Outcomes (PROs) | Week 12 and 24
Change from baseline in DAS28- CRP | Week 24
Safety and tolerability as indicated by adverse events, hematology, clinical chemistry, coagulation, urinalysis, electrocardiograms (ECGs) and vital signs | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ashrafzadeh, MD, FACR, Study Chair — Quintiles, Inc.
Locations (82):
- United States (31):
  - Vertex Investigational Site, Birmingham, Alabama
  - Vertex Investigational Site, Huntsville, Alabama
  - Vertex Investigational Site, Long Beach, California
  - Vertex Investigational Site, Tustin, California
  - Vertex Investigational Site, Boca Raton, Florida
  - Vertex Investigational Site, Daytona Beach, Florida
  - Vertex Investigational Site, New Port Richey, Florida
  - Vertex Investigational Site, North Miami Beach, Florida
  - Vertex Investigational Site, Ocala, Florida
  - Vertex Investigational Site, Tampa, Florida
  - Vertex Investigational Site, Springfield, Illinois
  - Vertex Investigational Site, Wichita, Kansas
  - Vertex Investigational Site, Kalamazoo, Michigan
  - Vertex Investigational Site, St Louis, Missouri
  - Vertex Investigational Site, Omaha, Nebraska
  - Vertex Investigational Site, Las Vegas, Nevada
  - Vertex Investigational Site, Clifton, New Jersey
  - Vertex Investigational Site, Freehold, New Jersey
  - Vertex Investigational Site, Brooklyn, New York
  - Vertex Investigational Site, Charlotte, North Carolina
  - Vertex Investigational Site, Durham, North Carolina
  - Vertex Investigational Site, Hickory, North Carolina
  - Vertex Investigational Site, Oklahoma City, Oklahoma
  - Vertex Investigational Site, Bethlehem, Pennsylvania
  - Vertex Investigational Site, Duncansville, Pennsylvania
  - Vertex Investigational Site, Jackson, Tennessee
  - Vertex Investigational Site, Austin, Texas
  - Vertex Investigational Site, Houston, Texas
  - Vertex Investigational Site, Mesquite, Texas
  - Vertex Investigational Site, San Antonio, Texas
  - Vertex Investigational Site, Clarksburg, West Virginia
- Argentina (2):
  - Vertex Investigational Site, Buenos Aires
  - Vertex Investigational Site, Santa Fe
- Bulgaria (4):
  - Vertex Investigational Site, Plovdiv
  - Vertex Investigational Site, Sevlievo
  - Vertex Investigational Site, Sofia
  - Vertex Investigational Site, Veliko Tarnovo
- Czechia (6):
  - Vertex Investigational Site, Brno
  - Vertex Investigational Site, Bruntál
  - Vertex Investigational Site, Mladá Boleslav
  - Vertex Investigational Site, Ostrava - Trebovice
  - Vertex Investigational Site, Prague
  - Vertex Investigational Site, Zlín
- Vertex Investigational Site, Tallinn, Estonia
- Germany (4):
  - Vertex Investigational Site, Cologne
  - Vertex Investigational Site, Leipzig
  - Vertex Investigational Site, Würzburg
  - Vertex Investigational Site, Zerbst
- Hungary (3):
  - Vertex Investigational Site, Baja
  - Vertex Investigational Site, Budapest
  - Vertex Investigational Site, Szikszó
- Mexico (4):
  - Vertex Investigational Site, Chihuahua City
  - Vertex Investigational Site, Cuauhtémoc
  - Vertex Investigational Site, San Luis Potos
  - Vertex Investigational Site, San Miguel Chapultepec
- Poland (7):
  - Vertex Investigational Site, Bialystok
  - Vertex Investigational Site, Elblag
  - Vertex Investigational Site, Krakow
  - Vertex Investigational Site, Lublin
  - Vertex Investigational Site, Poznan
  - Vertex Investigational Site, Torun
  - Vertex Investigational Site, Warsaw
- Romania (3):
  - Vertex Investigational Site, Brăila
  - Vertex Investigational Site, Bucharest
  - Vertex Investigational Site, Judetul Galati
- Russia (5):
  - Vertex Investigational Site, Kemerovo
  - Vertex Investigational Site, Moscow
  - Vertex Investigational Site, Ryazan
  - Vertex Investigational Site, Saint Petersburg
  - Vertex Investigational Site, Yaroslavl
- Serbia (3):
  - Vertex Investigational Site, Belgrade
  - Vertex Investigational Site, Niška Banja
  - Vertex Investigational Site, Novi Sad
- Slovakia (4):
  - Vertex Investigational Site, Bratislava
  - Vertex Investigational Site, Dunajská Streda
  - Vertex Investigational Site, Poprad
  - Vertex Investigational Site, Rimavská Sobota
- Ukraine (5):
  - Vertex Investigational Site, Donetsk
  - Vertex Investigational Site, Kharkiv
  - Vertex Investigational Site, Lviv
  - Vertex Investigational Site, Odesa
  - Vertex Investigational Site, Vinnytsia